CLINICAL TRIAL: NCT00317187
Title: Partially Blinded Study to Assess Reactogenicity & Safety of GSK Biologicals' Tritanrix™-HepB/Hib-MenAC vs Tritanrix™-HepB/Hiberix™ in Healthy Infants After a Hepatitis B Birth Dose
Brief Title: Safety Study of a Vaccine Against Meningitis in Infants (2,4 & 6 Months Age) After a Birth Dose of Hepatitis B.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 100791
Record Dates: First submitted 2006-02-17; First posted 2006-04-24 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis B; Diphtheria; Whole Cell Pertussis; Tetanus; Haemophilus Influenzae Type b
MeSH Terms: conditions — Hepatitis B; Diphtheria; Tetanus; Haemophilus Infections

ARMS (4):
- Hib-MenAC Lot 1 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 1 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hib-MenAC Lot 2 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 2 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hib-MenAC Lot 3 Group (Experimental): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB combined vaccine mixed extemporaneously with Meningitec conjugate vaccine Lot 3 at 2, 4 and 6 months of age as an intramuscular injections in the anterolateral part of the left thigh.
  Interventions: Biological: Tritanrix-HepB/Meningitec conjugate vaccine
- Hiberix Group (Active Comparator): Healthy male or female subjects aged 56 to 83 days of age at the time of the first study vaccine dose, with previous hepatitis B vaccine at birth, received Tritanrix-HepB vaccine mixed extemporaneously with conjugate vaccine Hiberix at 2, 4 and 6 months of age as intramuscular injection in the anterolateral part of the thigh.
  Interventions: Biological: Tritanrix/Hiberix vaccine

INTERVENTIONS:
Biological: Tritanrix-HepB/Meningitec conjugate vaccine — The full content of two monodose vials of Tritanrix-HepB vaccine vial was extracted and injected into the vial containing the lyophilized Meningitec (5/5/5) vaccine. The vial was agitated until the lyophilized vaccine pellet had completely dissolved. The reconstituted mixed vaccines were used promptly after reconstitution (within 30 minutes): one dose of 0.5 ml of the reconstituted Tritanrix- HepB/Meningitec vaccine was withdrawn from the vial and administered, the needle was changed before injection
  Other Names: DTPw-HBV/Hib-MenAC conjugate vaccine
  Arms: Hib-MenAC Lot 1 Group; Hib-MenAC Lot 2 Group; Hib-MenAC Lot 3 Group
Biological: Tritanrix/Hiberix vaccine — The full content of the Tritanrix-HepB vaccine vial was extracted and injected into the vial containing the lyophilized Hiberix vaccine. The vial was agitated until the lyophilized vaccine pellet had completely dissolved. The reconstituted mixed vaccines were used promptly after reconstitution (within 30 minutes): the full volume of the mixed vaccines was withdrawn from the vial, the needle was changed before injection.
  Other Names: DTPw-HBV/Hib vaccine
  Arms: Hiberix Group

SUMMARY:
The purpose of this study is to compare the reactogenicity & safety of Tritanrix™-HepB/Hib-MenAC vaccine to the international standard of care, Tritanrix™-HepB/Hiberix™.

DETAILED DESCRIPTION:
Randomized study with four groups to receive one of the following vaccination regimens after a dose of hepatitis B vaccine given at birth:

* One of the 3 lots of GSK Biologicals' Hib-MenAC mixed with GSK Biologicals' Tritanrix™-HepB (3 different groups)
* GSK Biologicals' Tritanrix™-HepB/Hiberix™

ELIGIBILITY:
Inclusion criteria:

• Healthy infants 56-83 days of age at the time of the first vaccine dose, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks & has received a birth dose of hepatitis B vaccine within the first 3 days of life.

Exclusion criteria:

* Any confirmed immunodeficient condition, based on medical history and physical examination.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine, or planned administration during the study period with the exception of oral polio vaccine (OPV).
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type b, and/or meningococcal disease.
* History of diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and/or meningococcal disease or known exposure to these diseases since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 56 Days to 83 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2004-06-08 (Actual); Primary Completion 2005-01-16 (Actual); Study Completion 2005-01-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 1 | Days 0-3 post dose 1
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 2 | Days 0-3 post dose 2
Occurrence of fever > 38.5°C(axillary) during the 4-day follow-up period after dose 3 | Days 0-3 post dose 3

SECONDARY OUTCOMES:
Occurrence of solicited symptoms other than fever >38.5°C (axillary) during the 4-day follow-up period after each dose | Days 0-3 after each dose
Occurrence of unsolicited symptoms during the 31-day follow-up period after each dose | Day 0-30 after each dose
Occurrence of serious adverse events during the entire study period | Day 0 up to Month 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

REFERENCES:
- [Derived] Kerdpanich A, Warachit B, Kosuwon P, Gatchalian SR, Watanaveeradej V, Borkird T, Kosalaraksa P, Han HH, Hutagalung Y, Boutriau D, Dobbelaere K. Primary vaccination with a new heptavalent DTPw-HBV/Hib-Neisseria meningitidis serogroups A and C combined vaccine is well tolerated. Int J Infect Dis. 2008 Jan;12(1):88-97. doi: 10.1016/j.ijid.2007.06.002. Epub 2007 Aug 22. PMID 17716936